CLINICAL TRIAL: NCT01142973
Title: Prognostic Role of Coronary Artery plaquEs in Patients With Suspected Coronary Artery Disease Using Multislice of Computed Tomography (PREDICT)
Brief Title: The Clinical Course of Coronary Artery Disease in Coronary Multidetector Computed Tomographic Angiogram
Acronym: PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Assistant professor, Inje university ILSAN paik hospital
Other Study IDs: mdksu-mdct-001
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Study Type: Observational Study Design: Observational Model: Defined Population Observational Model: Natural History Time Perspective: Longitudinal Time Perspective: Prospective

DETAILED DESCRIPTION:
The natural history of individual plaques is unknown and needs to be established. Multidetector computed tomography (MDCT) angiography is a useful noninvasive imaging modality for assessing coronary plaque. Using MDCT, the researchers prospectively investigate the relationship between the presence of coronary plaques and cardiovascular events

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected coronary artery disease

Exclusion Criteria:

* Irregular heart beat
* Known allergy towards the contrast agent
* Renal dysfunction
* Impossible breath-hold
* Acute coronary syndrome patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: present typical/atypical chest pain
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2005-09; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Major cardiovascular events | 1 years after the MDCT-scan
  Cardiovascular death, non-fatal MI, or any stroke

SECONDARY OUTCOMES:
all causes of hospitalization | 1 years after the MDCT-scan
  Requiring hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sung Uk Kwon, M.D., Principal Investigator — Inje univ. ilsan paik hospital
Locations (1):
- Ilsan Paik hospital, Goyang, South Korea

REFERENCES:
- [Derived] Kim JB, Rogers IS, Kwon SU. Presence of plaques predicts worse outcomes in multi-detector computed tomography in patients with stable chest pain syndrome. Int J Cardiol. 2014 May 15;173(3):570-2. doi: 10.1016/j.ijcard.2014.03.118. Epub 2014 Mar 21. No abstract available. PMID 24717325